CLINICAL TRIAL: NCT05005013
Title: A Teleheath tDCS Approach to Decrease Cannabis Use: Towards Reducing Multiple Sclerosis Disability
Brief Title: A Teleheath tDCS Approach to Decrease Cannabis Use
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-01028
Record Dates: First submitted 2021-08-12; First posted 2021-08-13 (Actual); Results first posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Cannabis Use Disorder; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Transcranial Direct Current Stimulation; Mindfulness

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tDCS + Mindfulness (Experimental)
  Interventions: Other: Transcranial Direct Current Stimulation (tDCS); Other: Mindfulness
- Sham tDCS + Mindfulness (Sham Comparator)
  Interventions: Other: Sham - Transcranial Direct Current Stimulation (tDCS); Other: Mindfulness

INTERVENTIONS:
Other: Transcranial Direct Current Stimulation (tDCS) — tDCS is noninvasive brain stimulation device that modulates brain activity by delivering a low-intensity electrical current (2.0 mA) through sponge electrodes placed on the scalp.
  Arms: Active tDCS + Mindfulness
Other: Sham - Transcranial Direct Current Stimulation (tDCS) — The tDCS device is programmed to mimic active tDCS.
  Arms: Sham tDCS + Mindfulness
Other: Mindfulness — Participants will follow an audio track for guided mindfulness during the stimulation.

SUMMARY:
The study aims to evaluate the effect of Dorsolateral Prefrontal Cortex (DLPFC) Transcranial Direct Current Stimulation (tDCS) in decreasing distress and cannabis use. 46 participants with Relapse Remitting Multiple Sclerosis (RRMS), Cannabis Use Disorder (CUD) and elevated distress (K10 score of 10-35) will be recruited.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 21-65 (inclusive)
2. Seeking treatment to reduce or discontinue current cannabis use (smoke/vape/ingest)
3. Current Cannabis Use Disorder per DSM-V (MINI for DSM-V)
4. K10 score 10-35, inclusive (mild to high moderate distress)
5. Definite MS diagnosis, relapsing remitting (RRMS) subtype
6. PDDS score 0-7 (mild to moderate neurological disability, established to be able to complete procedures)
7. All medications stable for ≥ 1 month prior to enrollment and throughout the trial
8. Ability to understand the informed consent process and provide consent to participate in the study
9. Stable and continuous access to internet service, email (WiFi "hotspot" to be provided if needed)
10. Ability to use mobile devices
11. Fluent in English language (due to outcomes validated in English versions only)
12. WRAT-4 score ≥ 85

Exclusion Criteria:

1. MS clinical relapse or use of high dose of steroids in the past month
2. Patients under medical marijuana use prescribed by a clinician
3. Alcohol, tobacco, or substance use disorder other than cannabis
4. Primary neurologic, psychiatric or other medical disorder other than MS (entry MD screening)
5. Currently meets DSM-V criteria for moderate or severe substance use disorder in the past 6 months for any psychoactive substance.
6. Meets DSM-V criteria for current panic disorder, obsessive-compulsive disorder, post-traumatic stress syndrome, bipolar affective disorder, schizophrenia, dissociate disorders, and any other psychotic disorder or organic mental disorder
7. Current suicidal ideation or deemed to be of potential risk of self-injury
8. History of traumatic brain injury
9. Seizure disorder or recent (<5 years) seizure history
10. Metal implants in the head or neck
11. Enrolled in group or individual therapy for substance use disorder concurrent to intervention
12. Any skin disorder or skin sensitive area near stimulation locations
13. Pregnant or breastfeeding

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2024-02-14 (Actual); Study Completion 2024-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leigh Charvet, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared upon reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will have access to the data upon reasonable request. Requests should be directed to leigh.charvet@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active tDCS + Mindfulness | Sham tDCS + Mindfulness
Started | 31 | 16
Completed | 22 | 13
Not Completed | 9 | 3
Not completed — Withdrawal by Subject | 5 | 1
Not completed — Lost to Follow-up | 3 | 1
Not completed — Ineligibility | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active tDCS + Mindfulness | Sham tDCS + Mindfulness | Total
Number analyzed (Participants) | 22 | 13 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (11) | 46.2 (8.8) | 45.7 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 13 | 35
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 3 | 9
  Not Hispanic or Latino | 16 | 9 | 25
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 5 | 16
  White | 9 | 6 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 22 | 13 | 35

OUTCOME MEASURES:

1. Primary Outcome: Change in Kessler Psychological Distress Scale (K10) Score
Description: K10 is a 10-item questionnaire intended to yield a global measure of distress based on questions about anxiety and depressive symptoms that a person has experienced in the most recent 4 week period. Each question is given a score between 1 (none of the time) to 5 (all of the time). The total score ranges from 10 to 50. People with scores < 20 are likely to be well, 20-24 are likely to have a mild mental disorder, 25-29 are likely to have moderate mental disorder, and > 30 are likely to have a severe mental disorder.
Time Frame: Baseline, End of Intervention (Week 4)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active tDCS + Mindfulness | Sham tDCS + Mindfulness
Number analyzed (Participants) | 22 | 13
score on a scale | 6.4 (6.1) | 4.5 (4.2)

2. Primary Outcome: Change in Positive and Negative Affect Schedule Score - Positive Affect (PANAS-PA)
Description: The PA subscale includes 10 items describing positive mood states (e.g., "enthusiastic," "interested," "proud"), each rated on a Likert scale from 1 ("very slightly or not at all") to 5 ("extremely"). The total score ranges from 5-50; higher scores indicate greater levels of positive affect, reflecting an individual's engagement, energy, and pleasurable involvement with the environment.
Time Frame: Baseline, End of Intervention (Week 4)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active tDCS + Mindfulness | Sham tDCS + Mindfulness
Number analyzed (Participants) | 22 | 13
score on a scale | -1.3 (8.3) | 1.53 (8.6)

3. Primary Outcome: Change in Positive and Negative Affect Schedule Score - Negative Affect (PANAS-NA)
Description: The NA subscale consists of 10 items representing negative mood states (e.g., "upset," "nervous," "hostile"), each rated on a 5-point Likert scale from 1 ("very slightly or not at all") to 5 ("extremely"). The total score ranges from 5-50; higher scores reflect greater levels of negative affect, capturing distress and unpleasurable engagement with the environment.
Time Frame: Baseline, End of Intervention (Week 4)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active tDCS + Mindfulness | Sham tDCS + Mindfulness
Number analyzed (Participants) | 22 | 13
score on a scale | -0.7 (5.2) | 3 (4.3)

4. Primary Outcome: Change in Marijuana Craving Questionnaire (MCQ-17) Score
Description: MCQ is a standardized measure assessing marijuana craving. Each statement is scored on a 7 point likert scale of 1 (strongly disagree) and 7 (strongly agree).
  Questions 1-7 measure compulsivity. Questions 8-11 measure emotionality. Questions 12-15 measure expectations. Questions 16-17 measure purposefulness. The total score is the average response score and ranges from 1-7; higher scored indicate greater levels of marijuana craving.
Time Frame: Baseline, End of Intervention (Week 4)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active tDCS + Mindfulness | Sham tDCS + Mindfulness
Number analyzed (Participants) | 22 | 13
score on a scale | 0.27 (9.5) | 0.8 (9.7)

5. Primary Outcome: Change in Cannabis Withdrawal Scale (CWS) Score
Description: The version of CWS used in the study asks about symptoms experienced over the last 24 hours and consists of 19 statements. For each statement, its negative impact on normal daily activities is rated on a likert scale from 0 (not at all) to 10 (extremely). The total score ranges from 0 to 190; higher scores indicate that symptoms are having a larger negative impact on normal daily activities.
Time Frame: Baseline, End of Intervention (Week 4)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active tDCS + Mindfulness | Sham tDCS + Mindfulness
Number analyzed (Participants) | 22 | 13
score on a scale | 27.1 (29.4) | 7 (17.7)

6. Primary Outcome: Change in Number of Weekly Sessions of Cannabis Use
Description: Self-reported measure.
Time Frame: Baseline, End of Intervention (Week 4)
Measure: Mean (Standard Deviation); unit: Sessions per week
Arm/Group | Active tDCS + Mindfulness | Sham tDCS + Mindfulness
Number analyzed (Participants) | 22 | 13
Sessions per week | 1.36 (2.7) | 0.54 (1.9)

7. Primary Outcome: Change in Number of Monthly Sessions of Cannabis Use
Description: Self-reported measure.
Time Frame: Baseline, End of Intervention (Week 4)
Measure: Mean (Standard Deviation); unit: Sessions per month
Arm/Group | Active tDCS + Mindfulness | Sham tDCS + Mindfulness
Number analyzed (Participants) | 21 | 12
Sessions per month | 5.5 (9.1) | 3.33 (6.4)

8. Secondary Outcome: Change in Kessler Psychological Distress Scale (K10) Score
Description: as for outcome 1
Time Frame: End of Intervention (Week 4), Month 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active tDCS + Mindfulness | Sham tDCS + Mindfulness
Number analyzed (Participants) | 21 | 12
score on a scale | 0.3 (4.3) | 1.33 (4.1)

9. Secondary Outcome: Change in Positive and Negative Affect Schedule Score - Positive Affect (PANAS-PA)
Description: as for outcome 2
Time Frame: End of Intervention (Week 4), Month 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active tDCS + Mindfulness | Sham tDCS + Mindfulness
Number analyzed (Participants) | 21 | 13
score on a scale | -1.2 (6.4) | -0.6 (5.1)

10. Secondary Outcome: Change in Positive and Negative Affect Schedule Score - Negative Affect (PANAS-NA)
Description: as for outcome 3
Time Frame: End of Intervention (Week 4), Month 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active tDCS + Mindfulness | Sham tDCS + Mindfulness
Number analyzed (Participants) | 21 | 13
score on a scale | 2.6 (6.4) | 1 (4.7)

11. Secondary Outcome: Change in Marijuana Craving Questionnaire (MCQ-17) Score
Description: as for outcome 4
Time Frame: End of Intervention (Week 4), Month 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active tDCS + Mindfulness | Sham tDCS + Mindfulness
Number analyzed (Participants) | 21 | 13
score on a scale | 2.66 (9.3) | 2.53 (9.6)

12. Secondary Outcome: Change in Cannabis Withdrawal Scale (CWS) Score
Description: as for outcome 5
Time Frame: End of Intervention (Week 4), Month 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active tDCS + Mindfulness | Sham tDCS + Mindfulness
Number analyzed (Participants) | 22 | 13
score on a scale | 8 (22) | 4.5 (29.4)

13. Secondary Outcome: Change in Number of Weekly Sessions of Cannabis Use
Description: Self-reported measure.
Time Frame: End of Intervention (Week 4), Month 3
Measure: Mean (Standard Deviation); unit: Sessions per week
Arm/Group | Active tDCS + Mindfulness | Sham tDCS + Mindfulness
Number analyzed (Participants) | 21 | 13
Sessions per week | 0.23 (2.1) | 0.5 (2.5)

14. Secondary Outcome: Change in Number of Monthly Sessions of Cannabis Use
Description: Self-reported measure.
Time Frame: End of Intervention (Week 4), Month 3
Measure: Mean (Standard Deviation); unit: Sessions per month
Arm/Group | Active tDCS + Mindfulness | Sham tDCS + Mindfulness
Number analyzed (Participants) | 20 | 13
Sessions per month | 1.7 (7.4) | 2.6 (10.1)

ADVERSE EVENTS:
Time Frame: 4 weeks
Description: non-systematic assessment: self-reporting by participants
Arm/Group | Active tDCS + Mindfulness | Sham tDCS + Mindfulness
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/13
Other Adverse Events (participants affected / at risk) | 0/22 | 1/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active tDCS + Mindfulness (N=22) | Sham tDCS + Mindfulness (N=13)
Minor skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-17): https://cdn.clinicaltrials.gov/large-docs/13/NCT05005013/Prot_SAP_001.pdf
  • Informed Consent Form (2023-10-17): https://cdn.clinicaltrials.gov/large-docs/13/NCT05005013/ICF_000.pdf